CLINICAL TRIAL: NCT05328219
Title: Effectiveness of Gum Chewing on Polyethylene Glycol (PEG) Related Intake Adherence, GI Side Effects and Bowel Preparation Among Patients Undergoing Colonoscopy
Brief Title: Effectiveness of Gum Chewing on Polyethylene Glycol Related Intake Adherence, GI Side Effects and Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ILBSIndia21
Record Dates: First submitted 2021-12-30; First posted 2022-04-14 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-01

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; Chewing gum; Intake Adherence; Bowel preparation
MeSH Terms: interventions — Chewing Gum; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing gums with PEG solution (Experimental): The investigator provide the chewing gums with PEG solution to the experimental group.
  Interventions: Other: Chewing gums with PEG solution
- Standard of Care (Active Comparator): Care provided as per the standard existing routine.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Chewing gums with PEG solution — Patients undergoing colonoscopy under experimental group was advised to take 2L of PEG solution and packets of sugarless sweet mint flavored chewing gums.
  The patients are advised to Chew one stick of sugarless gum for at least 10 min after taking each glass of PEG solution and discard the chewing gum before taking next glass.
  Arms: Chewing gums with PEG solution
Other: Standard of care — Standard of care
  Arms: Standard of Care

SUMMARY:
Problem statement An Experimental Study to assess the effectiveness of Gum Chewing on Polyethylene Glycol (PEG) Related Intake Adherence, GI Side Effects and Bowel Preparation among Patients Undergoing Colonoscopy at ILBS, New Delhi.

Objectives of the study

The objectives of the study are:

Primary objective

1. To compare the effect of gum chewing in experimental vs. control groups in terms of PEG Related Intake Adherence, GI side effects and Bowel Preparation among Patients Undergoing Colonoscopy.

Secondary objective

1. To find the relationship of total amount of fluid taken with GI side effects and Bowel Preparation variables in patients undergoing colonoscopy under experimental group.
2. To determine the association of PEG Related Intake Adherence, GI side effects and Bowel Preparation among Patients with socio-demographic and clinical variables in patients undergoing colonoscopy under experimental group.

DETAILED DESCRIPTION:
Aim of the study To evaluate the effectiveness of Gum Chewing on Polyethylene Glycol (PEG) Related Intake Adherence, GI Side Effects and Bowel Preparation among Patients Undergoing Colonoscopy at ILBS, New Delhi.

Operational Definitions

Assess:

In this study, Assess refers to evaluating the effectiveness of Gum Chewing on Polyethylene Glycol (PEG) Related Intake Adherence, GI Side Effects and Bowel Preparation among Patients Undergoing Colonoscopy at ILBS, New Delhi.

Effectiveness:

In this study, effectiveness refers to degree to which gum chewing is successful in improving the intake adherence, GI side effects and bowel preparation from taking PEG solution among patients undergoing colonoscopy in experimental group as compared with the control group.

Chewing gum:

In this study, commercially available sugar free chewing gum was used, these were made with a delicious sweet mint flavour for a clean and fresh feeling and chewing gum with the PEG solution was taken as per the evidenced based protocol.

Ingredients: Sorbitol, Gum Base, Glycerol, Natural and Artificial Flavors; Less than 2% of: Hydrogenated Starch Hydrolysate, Aspartame, Mannitol, Acesulfame K, Soy Lecithin, Xylitol, Colors (Blue 1 Lake, Beta-Carotene), BHT (To Maintain Freshness).

GI Side Effects:

In this study, GI side effects refers to occurrence of gastro intestinal symptoms including abdominal discomfort, nausea, vomiting and retching secondary to the intake of PEG solution for bowel preparation in patients undergoing colonoscopy.

Abdominal discomfort:

In this study, abdominal discomfort refers to the sense of bowel movement and abdominal pain caused by intake of polyethylene glycol solution assessed by Numerical Rating Scale.

Nausea, Vomiting and Retching:

In this study, Nausea was defined as the desire to vomit without indulging in expulsive muscular movements. Vomiting was defined as the oral expulsion of gastrointestinal contents, while retching was the attempt to vomit without expelling any material. All these three parameters was assessed by using Rhodes index of nausea, vomiting and retching.

Intake Adherence:

In this study, it refers to the degree to which the patients undergoing colonoscopy follows the instructions related to PEG solution intake for bowel preparation. It was measured in terms of the total amount of PEG solution ingested, the total time taken for ingestion, extra fluid taken and total fluid taken before the colonoscopy.

Bowel Preparation:

In this study, bowel preparation refers to the extent to which the colon was cleared off the fecal matter following PEG solution ingestion in the patient undergoing colonoscopy. It was assessed by the colonoscopist using BBPS.

Polyethylene glycol solution:

In this study, PEG solution was given for bowel preparation for patients undergoing colonoscopy as prescribed by doctors. It was available in form of packet i.e., to be dissolved in 2 L of water. Patient was instructed to ingest whole solution within 2 hours as per the ingestion protocol.

Patient:

In this study, patient refers to the individual who was advised for colonoscopy for therapeutic or diagnostic purpose during the data collection period at OPDs of ILBS.

Colonoscopy:

In this study, colonoscopy refers to the elective procedure done to examine the colon for diagnostic and/or therapeutic purposes of various diseases like colorectal cancer, intestinal obstruction, GI bleeding etc.

Development and Description of Tools

Tools were prepared on an extensive review of books, journals, articles, Guide and Expert's opinion and investigators personal experience.

For the selection and preparation of tools, the following steps were taken:

* Planning for required tools.
* An extensive review of tools used in various literatures was undertaken.
* Discussion with Guides, Peer group and Professionals.
* A formal observation in the concerned area of the study.
* Requirement of the tools according to objectives and the conceptual framework were sought.
* Opinion of 9 Experts was sought to determine the clarity, relevance, representativeness, comprehensiveness, ambiguity and simplicity of the tools.

Thus the most appropriate tools were used in the present study. These tools were majorly divided into six sections as follows:

Structured Questionnaires Section I: Subject Data Sheet which further consist of

* Section A- Socio-Demographic Variables
* Section B- Clinical Variables Section II: Intake adherence Standardized Tools Section III: Numerical Rating Scale Section IV: The Rhodes Index of Nausea, Vomiting and Retching (INVR). Section V: Boston Bowel Preparation Scale. Structured Tools Section VI: Record Sheets
* Patient's Log Book

ELIGIBILITY:
Inclusion Criteria:

* OPD Patients who -

  * Have been planned for elective colonoscopy for therapeutic and/or diagnostic purposes.
  * Have been prescribed PEG solution for bowel preparation.
  * Are able to chew gum.
  * Are willing to participate in the study.
  * Can read and write English or Hindi.

Exclusion Criteria:

* Patients who -

  * Are critically ill.
  * Are on anti-emetic therapy.
  * Have some psychiatric issues making them unable to follow the instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete intake of PEG solution (2 litre) in both groups | up to 5 weeks
  Intake Adherence among Patients Undergoing Colonoscopy was assessed by Intake Adherence tool comprises of 4 items which include time spent in ingesting the whole PEG solution in minutes, total amount of PEG solution taken, extra fluid taken other than PEG solution, total amount of fluid taken in milliliters.
Number of patients with change in GI side effects related to PEG solution in both groups | up to 5 weeks
  GI side effects among Patients Undergoing Colonoscopy was assessed by Numerical Rating Scale and the Rhodes Index of Nausea, Vomiting, And Retching (INVR).
Improvement in bowel preparation in both groups | up to 5 weeks
  Bowel Preparation among Patients Undergoing Colonoscopy was assessed by Boston Bowel Preparation Scale. A four-point scoring system with maximum score of 9 and minimum score of 0 applied to each of the three broad regions of the colon: the right colon (including the cecum and ascending colon), the transverse colon (including the hepatic and splenic flexures), and the left colon (including the descending colon, sigmoid colon, and rectum).

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Ms Chaudhary, Nursing, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Pooja Chaudhary, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No